CLINICAL TRIAL: NCT02250716
Title: A Comparison of Immediate Treatment of CIN1 With Cryotherapy and Regular 12 Month Cytology Follow up in HIV Seropositive Women
Brief Title: A Comparison of Immediate Treatment of CIN1 With Cryotherapy and 12 Month Cytology Follow up in HIV Seropositive Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Cynthia S Firnhaber, Associate Professor of Medicine, University of Witwatersrand, South Africa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIN1
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Cervical Dysplasia
Keywords: CIN1; HIV seropositive women; Cryotherapy
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Experimental): Immediate treatment with Cryotherapy and 12 month cytology and histology follow-up
  Interventions: Procedure: cryotherapy
- Arm 2 (No Intervention): 12 month cytology and histology follow-up

INTERVENTIONS:
Procedure: cryotherapy — cryotherapy for cervical intraepithelial neoplasia in HIV infected women vs control arm of standard of care (repeat pap smear in 1 year)
  Arms: Arm 1

SUMMARY:
Based on the high incidence of cervical cancer and high grade dysplasia and increased progression and incomplete treatment of CIN2 and 3 in South Africa, we propose to study the effect of cryotherapy among HIV-positive women diagnosed with CIN 1 versus regular 12 month cytology follow-up. This study will be a dual-arm, open-label, randomized clinical trial for HIV-infected women diagnosed with CIN 1 and receiving care at the Themba Lethu Clinic, Helen Joseph Hospital, Johannesburg, South Africa. CIN 1 will be identified from patients who have had a colposcopic biopsy for persistent LSIL as per standard of care.

DETAILED DESCRIPTION:
Women with HIV have a higher risk of cervical cancer. Screening and treatment formaly of the disease is limited die to poor access of screening programs and multiple visits. Women with HIV also have high progressions rates of disease amd my need to be treated earliers. Cryotherapy is a low option and very easy to implement especially in low resource provinces.

* It is cheaper and easier to administer than Large Loop electrosurgical excision procedure (LLETZ)
* No histology or transportation costs of specimens
* Less invasive than LLETZ
* It is nurse driven and easily learned
* It decreases loss to follow-up of patients due to reduced waiting time, transportation costs, time off work and HIV stigma

ELIGIBILITY:
Inclusion Criteria:

* HIV -infected women whose biopsy proves CIN1 and who consent to study participants and procedures
* CIN1 with no visible lesion
* The entire ectocervical lesion should cover less than 75% of the cervix and not more than 2 - 3mm into the endocervical canal

Exclusion Criteria:

* Pregnant women
* Known and previous treatment for HSIL by any method (Cryotherapy, LEEP or cone biopsy)
* Women who are menstruating or who have active pelvic inflammatory disease will be deferred from the study until the infection is cleared or the menstrual cycle has ended; the patient may then participate in the study.
* Unsatisfactory colposcopic examination defined as inability to see the extent of the lesion in the endocervical canal and lesions deemed ineligible for cryotherapy by an OB/GYN specialist.
* Previous hysterectomy with removal of the cervix

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Regresson of CIN1 to a normal biopsy | 12 month
  Treatment failure is the progression of CIN1 to CIN2

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia S Firnhaber, MD, Principal Investigator — University of Witwatersrand, South Africa
Locations (1):
- University of Witwatersrand/Helen Joseph Hospital, Johannesburg, South Africa